CLINICAL TRIAL: NCT02864667
Title: Reader Study for Image Quality of Cone Beam Breast CT System
Status: Completed | Type: Observational
Sponsor: Koning Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-02
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Koning Breast CT (KBCT) was approved by FDA PMA. The X-ray detector originally used in Koning Breast CT was PaxScan 4030CB. Recently, Koning Breast CT uses a modified X-ray detector PaxScan 4030MCT. The modified detector is essentially identical to the previous model except a different detector housing which allows a narrower dead-space between the active area and the top of the housing.

The benefit of the modified detector is that it allows Koning to modify the patient exam table, achieving a flatter surface in the center. The flatter surface will increase patient comfort and improve workflow.

Meanwhile, flatter surface may also affect patient positioning and the coverage of the breast. The adequacy of the overall image quality with the new table/detector should be verified by radiologists.

DETAILED DESCRIPTION:
Koning Breast CT (KBCT) was approved by FDA PMA. The X-ray detector originally used in Koning Breast CT was PaxScan 4030CB. Recently, Koning Breast CT uses a modified X-ray detector PaxScan 4030MCT. The modified detector is essentially identical to the previous model except a different detector housing which allows a narrower dead-space between the active area and the top of the housing.

The benefit of the modified detector is that it allows Koning to modify the patient exam table, achieving a flatter surface in the center. The flatter surface will increase patient comfort and improve workflow.

Meanwhile, flatter surface may also affect patient positioning and the coverage of the breast. The adequacy of the overall image quality with the new table/detector should be verified by radiologists.

Images from ten (10) female patients (cases) with different breast sizes will be evaluated by 3 independent board-certified, MQSA-qualified radiologists (readers). The images were acquired from a separate clinical trial using KBCT system with the new table/detector.

Two readers will independently evaluate the image quality of each case and choose to "accept" or "reject" the case. If there is a disagreement for a certain case, a third reader will independently evaluate that case and give the final result.

ELIGIBILITY:
Inclusion Criteria:

* Females at least 35 years of age of any ethnicity
* Had a mammogram, read as BIRADS 1 or 2 (group I) or BIRADS 4 or 5 (group II)
* Will undergo study imaging no later than four weeks from date of mammogram
* Is able to undergo informed consent
* Require diagnostic imaging

Exclusion Criteria:

* Pregnancy
* Lactation
* Subjects with physical limitations that may prohibit resting prone on the exam table, such as, but not limited to: frozen shoulder, recent heart surgery, pace maker
* Subjects who are unable to tolerate study constraints
* Subjects who are unable to tolerate study constraints
* Subjects who have received radiation treatments to the thorax for malignant and nonmalignant conditions, such as (but not limited to)
* Treatment for enlarged thymus gland as an infant
* Irradiation for benign breast conditions, including breast inflammation after giving birth
* Treatment for Hodgkin's disease
* Subjects who have participated in a prior breast clinical trial that gave additional radiation dose, such as an additional mammogram
* Subjects who have received large numbers of diagnostic x-ray examinations for monitoring of disease such as (but not limited to) Tuberculosis Severe scoliosis

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is reported that digital mammography has reject rate between 8% and 10% and positioning is the major reason of rejection [1]. In order to prove that the KBCT detector/table is able to provide correct position and sufficient image quality to achieve equal or lower rejection rate than mammography, a minimum number of 10 cases is required.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Rejection Rate | One hour training session followed by a one hour reading session

IPD SHARING:
Plan to Share IPD: No